CLINICAL TRIAL: NCT02476331
Title: A Randomized Control Trial of Cognitive Training in Euthymic Bipolar Disorder
Brief Title: A Trial of Cognitive Training in Euthymic Bipolar Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Student no longer enrolled in program.
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Vina M. Goghari, Dr., University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB14-0767
Record Dates: First submitted 2015-06-15; First posted 2015-06-19 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Bipolar Disorder
Keywords: Cognitive training; Working memory; Emotion regulation
MeSH Terms: conditions — Bipolar Disorder; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive training (Experimental): The neurocognitive training program will be provided by an online platform called BrainGymmer (https://www.braingymmer.com/en/brain-games/). The experimental group will complete the working memory training, which involves three games: N-back, Multi-Memory, and Moving Memory. These games are designed to engage processes involving updating and manipulation of information. All of the training games provided by BrainGymmer are adaptive, meaning that the level of difficulty increases as users develop expertise on a given task. Participants randomized to the cognitive training arm will complete the training games for 30 minutes per day, 5 days a week, for a total of 10 weeks.
  Interventions: Behavioral: Working memory training
- Control (No Intervention): The control group will wait 10-weeks, during which they will receive treatment-as-usual (TAU), which might involve pharmacotherapy, psychotherapy, or both. After the 10-week waiting period, participants will complete post-testing assessments.

INTERVENTIONS:
Behavioral: Working memory training — The neurocognitive training program will be provided by an online platform called BrainGymmer (https://www.braingymmer.com/en/brain-games/). The experimental group will complete the working memory training, which involves three games: N-back, Multi-Memory, and Moving Memory. These games are designed to engage processes involving updating and manipulation of information. All of the training games provided by BrainGymmer are adaptive, meaning that the level of difficulty increases as users develop expertise on a given task. Participants randomized to the cognitive training arm will complete the training games for 30 minutes per day, 5 days a week, for a total of 10 weeks.
  Arms: Cognitive training

SUMMARY:
Bipolar disorder (BD) is characterized by extreme changes in mood and emotion dysregulation. Mood changes are episodic in nature, with distinct periods of mania, depression, and asymptomatic periods of euthymia. In addition to impairments in mood, cognitive impairments are a common feature of the disorder. These cognitive impairments persist during periods of euthymia and are associated with negative clinical and psychosocial outcomes. Specifically, individuals with BD show impairments in executive functions. Recent studies show that emotion regulation can be down-regulated by taxing executive functions, and it can be improved with working memory training, a specific component of executive functions. These initial studies show that emotion regulation is under executive control in healthy individuals; however, the nature of this relationship is not well understood in populations that are affected by impairments in both executive control and emotion regulation. Previous work on cognitive training has not targeted specific cognitive domains with an emphasis on understanding the underlying mechanisms that promote change. Moreover, well-controlled randomized control trial (RCT) studies are needed in order to provide high quality evidence to inform the efficacy of cognitive training interventions for psychiatric populations. The aim of the proposed study is to use a commercially available cognitive training program to study the effects of working memory training on cognitive, clinical, and psychosocial outcomes in patients with BD. We hypothesize that training working memory will lead to improvements in cognitive and emotional functioning, leading to downstream changes that will positively impact untrained outcomes, such as mood and community functioning.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18 and 65 years
* Clinically diagnosed with bipolar disorder I or bipolar disorder II and currently in a euthymic state
* Normal, or corrected to normal, vision and hearing
* Able to provide informed consent

Exclusion Criteria:

* Meeting Diagnostic and Statistical Manual 5th edition (DSM-5) diagnostic criteria for a current major depressive episode, manic episode, or hypomanic episode
* Past electroconvulsive therapy (ECT)
* Past Transcranial Magnetic Stimulation therapy (TMS)
* Past 3 month history of substance abuse
* Diagnosed with a medical condition known to affect cognition (e.g., endocrine disease)
* Score less than 70 on the Wechsler Abbreviated Scale of Intelligence (WASI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Working memory capacity | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the Automated Operation Span task (AOSPAN), Wechsler Adult Intelligence Scale (WAIS-IV) Digit Span and Maintenance and Manipulation task
Emotion regulation | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the Emotional Stroop task and Emotional N-back task
Fluid intelligence | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the Raven's Progressive Matrices (RPM) task

SECONDARY OUTCOMES:
Depression symptom severity | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the 17-item Hamilton Rating Scale for Depression (HRDS-17)
Manic symptom severity | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the Young Mania Rating Scale (YMRS)
Community functioning | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the Functioning Assessment Short Test (FAST)

OTHER OUTCOMES:
Decision making and impulsivity | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the Delay Discounting Task
Executive functioning: inhibition and set shifting | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with the Delis-Kaplan Executive Functions System (D-KEFS) Color-Word Interference Test
Executive functioning: categorization and set-shifting | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with D-KEFS Sorting Test
Theory of mind reasoning | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Hinting Task
Motivation | Throughout the 10 weeks of training
  Measured with the Intrinsic Motivation Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Vina Goghari, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] Lawlor-Savage L, Goghari VM. Working memory training in schizophrenia and healthy populations. Behav Sci (Basel). 2014 Sep 3;4(3):301-319. doi: 10.3390/bs4030301. eCollection 2014 Sep. PMID 25379283